CLINICAL TRIAL: NCT03811691
Title: Clinical Investigation of ENO/TEO/OTO Pacing System Under MRI Environment
Acronym: CAPRI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IBSY06 - CAPRI
Record Dates: First submitted 2019-01-15; First posted 2019-01-22 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Intervention Model Description: This study is an interventional, prospective, multicenter, open label, two arms parallel non-comparative non-randomized study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.5 Tesla MRI Scan (Other): Subjects will undergo 1.5T MRI exam
  Interventions: Diagnostic Test: MRI exam
- 3 Tesla MRI Scan (Other): Subjects will undergo 3T MRI exam
  Interventions: Diagnostic Test: MRI exam

INTERVENTIONS:
Diagnostic Test: MRI exam — Pacing system safety and stability under MRI scan environment

SUMMARY:
The interest of the CAPRI study is to confirm the safety and the efficacy of the ENO/TEO/OTO pacing system when used under 1.5 or 3 Tesla MRI environment and in accordance with the MRI solutions guideline.

DETAILED DESCRIPTION:
The purpose of CAPRI study is to confirm the safety and the efficacy of the CE marked MR conditional pacing system composed of the ENO, TEO or OTO pacemaker with VEGA pacing lead(s). Conditions to undergo an MRI scan are provided in the MRI solutions guideline.

The primary objective is to confirm the clinical safety of the ENO/TEO/OTO pacing system when used under 1.5 and 3 Tesla specific MRI conditions without scan exclusion zone.

The study secondary main objectives are aiming to assess the performance of the MR conditional pacing system in the right atrium and ventricle at 1 month following the MRI scan:

* Stability of the Pacing Capture Threshold
* Stability of the lead sensed amplitude

ELIGIBILITY:
Inclusion Criteria:

Subjects who meet all the following criteria at the time of inclusion visit may be included:

* Already implanted in the left or right pectoral region for at least 6 weeks with:

  * ENO, TEO or OTO single chamber rate response (SR) pacemaker with a VEGA pacing lead, or
  * ENO, TEO or OTO dual chamber rate response (DR) pacemaker with two VEGA pacing leads.
* Implanted pacing system must fulfill the following parameters:

  * Battery impedance is < 5 Kilo Ohm (kΩ)
  * Pacing capture threshold value is ≤ 2 Volts (V) at 0.35 millisecond (ms)
  * Lead impedance value between 200Ω and 3000Ω
  * No diaphragmatic or pectoral stimulation at 5V/1ms
  * P-wave minimum sensed amplitude ≥ 1mV for patients with sinus rhythm
  * R-wave minimum sensed amplitude ≥ 4mV for patients with spontaneous conduction rhythm
* Must agree to undergo a non clinically-indicated MRI scan without intravenous injection and without sedation;
* Have reviewed, signed and dated informed consent.

Subjects who meet any of the following criteria are not eligible to be included in the study:

* Included in another clinical study that could confound the results of this study such as studies involving intra-cardiac device;
* Have other active or abandoned cardiac implants already implanted;
* Have other active or passive non MR conditional devices implanted such as metallic foreign body;
* Have a history of brain aneurysm with ferromagnetic clipping;
* Have a planned cardiac surgery within the 3 months of inclusion;
* Have a medical MRI examination prescription planned within the 3 months of inclusion;
* Age less than 18 years old or under guardianship or kept in detention;
* Known pregnancy, women breastfeeding or in childbearing age without an adequate contraceptive method ;
* Be unavailable for the scheduled follow-up associated with this clinical study or refusal to cooperate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Freedom from MRI-related complications following the MRI scan of the ENO/TEO/OTO pacing system | 1 month post MRI
  An MRI-related complication is defined as a Serious Adverse Event (SAE) that led to death or to an invasive intervention or a Device Deficiency that causes the termination of any significant device function per Clinical Event Committee (CEC) adjudication.
  The primary endpoint will be assessed independently for each arm of the study (1.5 and 3 Tesla MRI scan).

SECONDARY OUTCOMES:
Ventricular Pacing Capture Threshold (PCT) stability in the right atrium and ventricle following the MRI scan | 1 month post MRI
  Subject's ventricular pacing capture threshold will be measured in Volt (V) at 0.5ms at baseline (at the MRI visit - just before the MRI scan) and at 1 month Post-MRI visit. A success is defined as a PCT increase less than or equal to 0.5V at 0.5ms between the two visits. The secondary endpoints will be assessed independently for each arm of the study (1.5 and 3 Tesla MRI scan).
Atrial Pacing Capture Threshold stability in the right atrium and ventricle following the MRI scan | 1 month post MRI
  Subject's atrial pacing capture threshold will be measured in Volt (V) at 0.5ms at Baseline (at the MRI visit - just before the MRI scan) and at 1 month Post-MRI visit. A success is defined as a PCT increase less than or equal to 0.5V at 0.5ms between the two visits. The secondary endpoints will be assessed independently for each arm of the study (1.5 and 3 Tesla MRI scan).
Ventricular sensed amplitude stability in the right atrium and ventricle following the MRI scan | 1 month post MRI
  Subject's ventricular minimum sensed amplitude will be measured in mV at Baseline (at the MRI visit - just before the MRI scan) and at 1 month Post-MRI visit. A success is defined as 50% or less decrease between the two visits. If subject's ventricular minimum sensed amplitude is less or equal to 4mV at time of baseline, then this subject will not count for this endpoint. The secondary endpoints will be assessed independently for each arm of the study (1.5 and 3 Tesla MRI scan).
Atrial sensed amplitude stability in the right atrium and ventricle following the MRI scan | 1 month post MRI
  Subject's atrial minimum sensed amplitude will be measured in mV at baseline. A success is defined as 50% or less decrease between the two visits. If subject's atrial minimum sensed amplitude is less or equal to 1mV at time of Baseline (at the MRI visit - just before the MRI scan) and at 1 month Post-MRI visit, then this subject will not count for this endpoint.The secondary endpoints will be assessed independently for each arm of the study (1.5 and 3 Tesla MRI scan).

CONTACTS AND LOCATIONS:
Locations (1):
- MicroPort CRM, Clamart, Haut de Seine, France

IPD SHARING:
Plan to Share IPD: No